CLINICAL TRIAL: NCT00973453
Title: Dose Tolerability Study With High Dose PURETHAL Mites in Allergic Rhinitis / Rhinoconjunctivitis Patients
Brief Title: Study With High Dose PURETHAL Mites in Allergic Rhinitis/Rhinoconjunctivitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PM/0028
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: non-seasonal allergy; house dust mite; immunotherapy; dose tolerability
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Slow regimen (Other)
  Interventions: Drug: PURETHAL Mites 20,000 AUeq/ml
- Intermediate regimen (Other)
  Interventions: Drug: PURETHAL Mites 20,000 AUeq/ml
- Fast regimen (Other)
  Interventions: Drug: PURETHAL Mites 20,000 AUeq/ml

INTERVENTIONS:
Drug: PURETHAL Mites 20,000 AUeq/ml — Group 1: slow regimen (12+2 injections) Initial treatment: incremental weekly dose of 0.05, 0.1, 0.2, 0.3, 0.4, 0.5, 0.6, 0.8, 1.0, 1.2*, 1.6* and 2.0* ml Additional maintenance: 2 two-weekly injections 2.0* ml
  *Injection volumes larger than 1 ml will be given as 2 separate injections of equal volume within an area of 1 cm.
  Other Names: Immunotherapy for house dust mites allergy
  Arms: Slow regimen
Drug: PURETHAL Mites 20,000 AUeq/ml — Group 2: intermediate regimen (9+2 injections) Initial treatment: incremental weekly dose of 0.1, 0.2, 0.4, 0.6, 0.8, 1.0, 1.2*, 1.6* and 2.0* ml.
  Additional maintenance: 2 two-weekly injections 2.0* ml
  *Injection volumes larger than 1 ml will be given as 2 separate injections of equal volume within an area of 1 cm.
  Other Names: Immunotherapy for house dust mites allergy
  Arms: Intermediate regimen
Drug: PURETHAL Mites 20,000 AUeq/ml — Group 3: fast initial treatment (6+2 injections) Initial treatment: incremental weekly dose of 0.2, 0.4, 0.8, 1.2*, 1.6* and 2.0*ml.
  Additional maintenance: 2 two-weekly injections 2.0* ml
  *Injection volumes larger than 1 ml will be given as 2 separate injections of equal volume within an area of 1 cm.
  Other Names: Immunotherapy for house dust mites allergy
  Arms: Fast regimen

SUMMARY:
The aim of the study is to establish the maximum tolerated dose of PURETHAL Mites that is achieved by 90% of the patients with less than 20% of the injections giving rise to a swelling of > 5 cm and the optimal regimen to reach this maximum dose will be determined.

DETAILED DESCRIPTION:
The tolerability and safety of three different initial treatment regimens PURETHAL mites in patients with allergic rhinitis / rhinoconjunctivitis induced by house dust mites will be evaluated and the optimal regimen to reach the maximum tolerated dose will be determined. The maximum intended dose is a 4-fold dosage compared to the currently used maintenance dose of PURETHAL Mites. The tolerability and safety of the injections will be examined by means of determining the early and late local and systemic reactions. In addition, short-term efficacy of this high dose PURETHAL mites will be determined by means of the Clinical index score (CIS) and two surrogate efficacy markers; the conjunctival provocation test (CPT) and serum levels of allergen specific immunoglobulins (IgG and IgE). These efficacy parameters are purely indicative and not decisive for the further clinical development of PURETHAL Mites.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with perennial rhinitis or rhinoconjunctivitis, with or without mild asthma (FEV1 > 70%) for at least 2 years. with allergic symptoms related to HDM
2. Positive CPT test to HDM Der p, dose ≤10,000 AUeq/ml
3. Positive SPT to HDM Der p or Der f (mean wheal diameter ≥ 3mm)
4. Specific serum IgE-test (ssIgE > 0.7 U/ml) for HDM
5. Age ≥ 18 years
6. Written informed consent given

Exclusion Criteria:

1. Patients with concomitant sensitization i.e. positive SPT (mean wheal diameter ≥ 3 mm) to other allergens than HDM should not be included if they have clinical symptoms at the time of inclusion, related to the other allergen
2. Patients sensitized to pets should not be included if they live together with these pets or have clinical symptoms
3. Immunotherapy (including sublingual) with HDM within the last 5 years
4. Immunotherapy (including sublingual) during the study period
5. Chronic asthma or emphysema, particularly with a FEV1 ≤ 70% of predicted value or use of inhalation corticosteroids
6. Serious immuno-pathologic diseases or malignancies (including auto-immune diseases, tuberculosis)
7. Symptomatic coronary heart diseases or severe (even under treatment) arterial hypertension
8. Diseases with a contra-indication for the use of adrenaline
9. Patients who are using other aluminium preparations, e.g. antacids
10. Severe kidney disease
11. Use of systemic steroids
12. Treatment with systemic and local Beta-blockers or immunosuppressive drugs
13. Active infection of the target organs (nose or eyes)
14. Severe atopic dermatitis in case systemic immunosuppressive medication is used
15. Participation in a clinical study with a new investigational drug within the last 3 months
16. Pregnancy, lactation or inadequate contraceptive measures (adequate contraceptive measures will be the use of a contraceptive device or -pill)
17. Alcohol- or drug abuse
18. Lack of co-operation or severe psychological disorders
19. Institutionalisation by official or judicial order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Early Local Reactions (ELR) occurring 15 minutes after injection. Less than 20% of the injections should give rise to swelling at the injection site of > 5 cm in diameter occurring 15 minutes after injection. | 17, 14 or 11 weeks per patient for the respective groups

SECONDARY OUTCOMES:
Late Local Reactions (LLR) occurring within 24 hours after injection, and systemic reactions (SR). General adverse events will be recorded during complete study period. | 17, 14 or 11 weeks per patient for the respective groups
Clinical index score (CIS) during the study compared to baseline score (before treatment). | weekly during per patient treatment periods of 17, 14 or 11 weeks for the respective groups
Conjunctival provocation test one week after reaching 10,000 AUeq, 20,000 AUeq, or 40,000 AUeq for the respective groups compared to baseline. | after 7 weeks of treatment
Conjunctival provocation test 2 weeks after the patients have received two maintenance dosages compared to baseline score. | 17, 14 or 11 weeks for the respective treatment groups
Specific IgE and IgG measured 2 weeks after the patients have received two maintenance dosages compared to baseline score. | 17, 14 or 11 weeks for the respective treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Kleine-Tebbe, MD, Study Chair — UZDAA, Untersuchungszentrum Dermatologie, Allergologie und Asthma, Berlin, Germany
Locations (6):
- Germany (6):
  - Allergie-Centrum Charité, Klinik für Dermatologie, Venerologie und Allergologie, Charité Campus Mitte, Universitätsmedizin Berlin, Berlin
  - Hals, Nasen- und Ohrenheilkunde, Berlin
  - Allergy & Asthma Center Westend, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Allergologie HNO-Heilkunde, Schorndorf
  - Klinik für Dermatologie und Allergie, Krankenhaus Bad Cannstatt, Stuttgart